CLINICAL TRIAL: NCT01701765
Title: Epidemiological Study on Outcomes and Discharges of Psychiatric Patients Living in Italian Residential Facilities (PERDOVE)
Brief Title: Outcomes and Discharge of Long-stay Psychiatric Patients
Acronym: PERDOVE
Status: Completed | Type: Observational
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Giovanni de Girolamo, M.D., M.D., IRCCS Centro San Giovanni di Dio Fatebenefratelli
Other Study IDs: 2012-2-PEV
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Mental Disorders
Keywords: Severe mental disorders; Discharge; Outcome evaluation
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients in residential facilities: All patients staying in September 2010 in 23 medium-long term RFs of the St John of God Order in Northern Italy with a primary psychiatric diagnosis and younger than 65 years recruited.

SUMMARY:
An increasing number of severely ill patients require long-term care in non-hospital Residential Facilities (RFs). Despite the magnitude of this development, only a few detailed longitudinal studies on fairly larger samples of residents have provided important information about this population. The PERDOVE study is the first study carried out in Italy aimed at obtaining comprehensive data about the course and outcome of patients living in RFs, and test whether discharge to independent accommodations is a real option for many patients. The major aims are three: (1) to describe the sociodemographic, clinical, and treatment-related characteristics of patients treated in RFs during an index period in 2010; (2) to identify predictors, and characteristics associated to discharge at 1-year follow-up; and (3) to evaluate clinicians' predictions about the likelihood of home discharge for each individual patient. The primary endpoint was discharge within one year as a measure of good outcome. The PERDOVE study is an observational cohort study, involving 23 RFs all belonging to the St John of God Order, located in Northern Italy. The first step involves the evaluation of all RFs with a Structure Schedule, which assesses the following areas: logistics structure, general organization: internal rules, meals, clothing and personal hygiene; staff and users' characteristics and meetings, documentation system and evaluation activities; rehabilitative activities provided inside the RF itself. In the second step a research assistant completed a standardised assessment of each resident with the manager and staff; clinical diagnoses were made by treating clinicians. A number of standardised instruments were administered. At one year follow-up, changes in clinical and life conditions of the patients were evaluated and selected rating scales were administered again. For patients discharged to the community or to other RFs, a research assistant contacted the patient's psychiatrist and asked him/her to fill out the follow-up documentation. With regard to residents' discharge, investigators hypothesised that the likelihood of community discharge would be associated both with the level of social support outside the facilities, and with the degree of patients' psychological and social impairment.

ELIGIBILITY:
Inclusion Criteria:

* psychiatric diagnosis
* age < 65
* staying in september 2010 in any of 23 RFs located in Northern Italy

Exclusion Criteria:

* elderly patients (over 65 yrs)
* primary diagnosis of organic mental disorder
* refusal of signing an informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric patients staying in residential facilities.
Sampling Method: Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Discharge | 1 year
  Percentage of patients discharged home one year after the baseline assessment compared to patients staying in the same residential facility or transferred to other institutions (e.g., other residential facilities, nursing homes, jails, etc)

SECONDARY OUTCOMES:
Scores of standardized rating scales | 1 year
  Clinical psychopathology (BPRS), psychosocial functioning (PSP, HONOS, SLOF), Quality of life (WHOQOL, WHOQOL-SRPB, SWBS), physical conditions (PHI)
Satisfaction assessed with the VSSS | 1 year
  Satisfaction with the treatment received assessed with the Verona Service Satisfaction Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni de Girolamo, M.D., Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (4):
- Italy (4):
  - IRCCS Centro san Giovanni di Dio, Brescia, Brescia
  - IRCSS Sant'Ambrogio, Cernusco sul Naviglio, Milano
  - IRCCS Sacro Cuore di Gesù, San Colombano al Lambro, Milano
  - IRCCS Presidio Ospedaliero Beata Verigine della Consolata, San Maurizio Canavese, Torino

REFERENCES:
- [Derived] Lanfredi M, Candini V, Buizza C, Ferrari C, Boero ME, Giobbio GM, Goldschmidt N, Greppo S, Iozzino L, Maggi P, Melegari A, Pasqualetti P, Rossi G, de Girolamo G; PERDOVE group. The effect of service satisfaction and spiritual well-being on the quality of life of patients with schizophrenia. Psychiatry Res. 2014 May 15;216(2):185-91. doi: 10.1016/j.psychres.2014.01.045. Epub 2014 Feb 6. PMID 24582503
- [Derived] de Girolamo G, Candini V, Buizza C, Ferrari C, Boero ME, Giobbio GM, Goldschmidt N, Greppo S, Iozzino L, Maggi P, Melegari A, Pasqualetti P, Rossi G. Is psychiatric residential facility discharge possible and predictable? A multivariate analytical approach applied to a prospective study in Italy. Soc Psychiatry Psychiatr Epidemiol. 2014 Jan;49(1):157-67. doi: 10.1007/s00127-013-0705-z. Epub 2013 May 28. PMID 23712514
- See also: website of the coordinating centre — http://www.irccs-fatebenefratelli.it/sito/pagine/fatebenefratelli.php